CLINICAL TRIAL: NCT03526042
Title: Angiotensin-II Receptor Antibody Blockade With Losartan in Patients With Lupus Nephritis
Brief Title: Angiotensin-II Receptor Antibodies Blockade With Losartan in Patients With Lupus Nephritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Luis Eduardo Morales Buenrostro, Clinical Professor of Nephrology, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMM-1816,16/16-1
Record Dates: First submitted 2018-04-16; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Atherosclerosis; Lupus Nephritis
MeSH Terms: conditions — Atherosclerosis; Lupus Nephritis | interventions — Losartan; Angiotensin Receptor Antagonists; Enalapril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Intervention Model Description: Open randomized clinical trial with parallel group comparing AT1R-ab blockade with losartan and enalapril as a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan (Experimental): AT1R-ab effect can be blocked with the use of angiotensin-II receptor blockers. The participants will receive losartan.
  Interventions: Drug: Losartan
- Enalapril (Active Comparator): Angiotensin converting enzyme inhibitors are indicated in the management of active lupus nephritis but do not block the effect of AT1R-Ab.
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Losartan — Competitive blockade of AT1R-antibodies effect by binding to the angiotensin 1 receptor
  Other Names: Angiotensin receptor blocker
  Arms: Losartan
Drug: Enalapril — Renin-angiotensin-aldosterone system (RAAS) blockade without any effect on AT1R-antibodies effect or concentration (control group)
  Other Names: Angiotensin Converting Enzyme Inhibitor
  Arms: Enalapril

SUMMARY:
Antibodies directed against angiotensin-II receptor (AT1-Ab) are agonist antibodies previously studied in human diseases such as preeclampsia, transplantation and scleroderma. They act by binding to the AT1 receptor and their effects can be blocked with the use of angiotensin receptor blockers (ARB). In this randomized open clinical trial the investigators will study the effect of the blockade of AT1-Ab with losartan in carotid intima-media thickness progression in patients with lupus nephritis compared to patients treated with enalapril.

DETAILED DESCRIPTION:
Angiotensin-II type 1 receptor antibodies (AT1R-Ab) are agonist antibodies directed against the second loop of the AT1 receptor. These antibodies have been studied in human diseases such as preeclampsia, transplantation and scleroderma. A previous study from the investigators' group found an elevated prevalence of AT1R-Ab in patients with lupus nephritis. As these antibodies have been linked to atherosclerosis development this open randomized clinical trial was designed to evaluate the effect of AT1R-Ab blockade with losartan compared to the use of enalapril in the progression of carotid intima-media thickness (CIMT) in patients with active lupus nephritis.

Biopsy-proven lupus nephritis patients who tested positive for AT1R-Ab will be performed a CIMT measurement by Doppler ultrasound at the time of the biopsy and then at 12-months follow up.

The primary outcome will be the change in the CIMT in the course of 12 months in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form for the study
* Biopsy-proven lupus nephritis with proteinuria > 1.5g/g by 24 hour urine protein to creatinine ratio
* Need for immunosuppressive induction to remission therapy according to the treatment physician
* Systemic lupus erythematosus diagnosis based on at least 4 American College of Rheumatology criteria
* Age between 16 and 50 years

Exclusion Criteria:

* Patient does not want to participate in the study
* Comorbid disease such as diabetes mellitus with macro/microangiopathy, previous diagnosis of hypertension >5 years, scleroderma
* Comorbid findings in the histopathological analysis of the renal biopsy

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Carotid intima-media thickness change after 12 months of the intervention | 12 months
  Change in carotid intima-media thickness from baseline thickness at study entry to 12 months of follow up measured by Doppler ultrasound

SECONDARY OUTCOMES:
Response to treatment | 12 months
  Response to immunosuppressive treatment at 12 months
Arterial pressure | 12months
  Arterial pressure control recorded by 24-hour ambulatory blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Morales-Buenrostro, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03526042/Prot_SAP_000.pdf